CLINICAL TRIAL: NCT03840616
Title: Phase 3, Randomized, Double-Blind Study to Evaluate Efficacy and Safety of Oteseconazole (VT-1161) Oral Capsules vs Fluconazole and Placebo in Treatment of Acute Vulvovaginal Candidiasis in Subjects With Recurrent Vulvovaginal Candidiasis
Brief Title: Study of Oral Oteseconazole (VT-1161) for Acute Yeast Infections in Patients With Recurrent Yeast Infections
Acronym: ultraVIOLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mycovia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-017
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oteseconazole (VT-1161) 150mg capsule (Experimental): 600mg oteseconazole administered on Day 1 and 450mg administered on Day 2, followed by 150mg administered once weekly for 11 weeks staring on Day 14
  Interventions: Drug: Oteseconazole (VT-1161) 150mg capsule
- Fluconazole 150mg capsule / Placebo (Active Comparator): 150mg fluconazole administered every 72 hours in 3 sequential doses starting on Day 1, followed by placebo administered once weekly starting on Day 14
  Interventions: Drug: Fluconazole 150mg capsule; Drug: Placebo

INTERVENTIONS:
Drug: Oteseconazole (VT-1161) 150mg capsule — 600mg administered on Day 1 and 450mg administered on Day 2, followed by 150mg administered once weekly for 11 weeks staring on Day 14.
  Arms: Oteseconazole (VT-1161) 150mg capsule
Drug: Fluconazole 150mg capsule — 150mg administered every 72 hours in 3 sequential doses starting on Day 1.
  Arms: Fluconazole 150mg capsule / Placebo
Drug: Placebo — Administered once weekly starting on Day 14.
  Arms: Fluconazole 150mg capsule / Placebo

SUMMARY:
Recurrent vulvovaginal candidiasis (RVVC), also known as recurrent yeast infections, is defined as at least 3 episodes of acute vulvovaginal candidiasis (VVC) in the past 12 months. Several properties of oteseconazole (VT-1161) suggest it might be a safer and more effective treatment of RVVC than other oral antifungal medications.

This study will evaluate the effectiveness and safety of oteseconazole (VT-1161) for the treatment of acute VVC episodes in patients with RVVC and consists of 2 parts. The first part of the study is a 2-week induction phase for the treatment of the patient's current VVC episode when the patient will take either fluconazole or oteseconazole (VT-1161) according to a random assignment. The second part consists of an 11-week maintenance phase, when the patient will take either oteseconazole (VT-1161) or a placebo according to the random assignment from the first part of the study, and then a 37-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 3 or more episodes of acute VVC in the past 12 months
* Positive KOH test
* Total vulvovaginal signs and symptoms score of ≥3 at screening visit
* Total vulvovaginal signs and symptoms score of <3 at Day 14
* Must be able to swallow pills

Exclusion Criteria:

* Presence or a history of another vaginal or vulvar condition(s)
* Evidence of major organ system disease
* History of cervical cancer
* Poorly controlled diabetes mellitus
* Pregnant
* Recent use of topical or systemic antifungal or antibacterial drugs
* Recent use of immunosuppressive or systemic corticosteroid therapies

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - 34, Tucson, Arizona
  - 39, Encino, California
  - 25, Los Angeles, California
  - 22, Englewood, Colorado
  - 49, Boca Raton, Florida
  - 14, Gainesville, Florida
  - 13, Leesburg, Florida
  - 33, Loxahatchee Groves, Florida
  - 36, Miami, Florida
  - 17, Savannah, Georgia
  - 27, Idaho Falls, Idaho
  - 10, Nampa, Idaho
  - 62, Chicago, Illinois
  - 41, Fort Wayne, Indiana
  - 30, Marrero, Louisiana
  - 50, Dearborn Heights, Michigan
  - 29, Saginaw, Michigan
  - 55, Traverse City, Michigan
  - 32, Troy, Michigan
  - 26, Kansas City, Missouri
  - 42, New Brunswick, New Jersey
  - 47, Ocean City, New Jersey
  - 37, Charlotte, North Carolina
  - 38, Fayetteville, North Carolina
  - 15, Columbus, Ohio
  - 18, Bluffton, South Carolina
  - 48, Myrtle Beach, South Carolina
  - 20, Bristol, Tennessee
  - 21, Murfreesboro, Tennessee
  - 24, Austin, Texas
  - 23, Fort Worth, Texas
  - 63, Katy, Texas
  - 58, League City, Texas

REFERENCES:
- [Derived] Vanreppelen G, Nysten J, Baldewijns S, Sillen M, Donders G, Van Dijck P. Oteseconazole (VIVOJA) for prevention of recurrent vulvovaginal candidiasis. Trends Pharmacol Sci. 2023 Jan;44(1):64-65. doi: 10.1016/j.tips.2022.10.004. Epub 2022 Nov 14. No abstract available. PMID 36396498

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After providing consent, 251 subjects were screened and, of those, a total of 219 subjects were randomly assigned to the oteseconazole or fluconazole/placebo group for a 2-week induction phase. During the induction phase, subjects received either oteseconazole or fluconazole. Subjects whose presenting acute VVC episode resolved during the induction phase (a total of 185 subjects) entered a 48-week maintenance phase comprised of an 11-week treatment period and a 37-week follow-up period.
Pre-assignment Details: Of the 251 subjects screened, 32 did not meet eligibility requirements and were not enrolled (i.e., not assigned to a treatment arm for the 2-week induction phase).
Groups:
- Oteseconazole (VT-1161): 600mg on Day 1 and 450mg on Day 2, followed by 150mg once weekly for 11 weeks starting on Day 14.
- Fluconazole / Placebo: 150mg fluconazole every 72 hours in 3 sequential doses starting on Day 1, followed by placebo once weekly for 11 weeks starting on Day 14.
Period: 2-Week Induction Phase
Arm/Group | Oteseconazole (VT-1161) | Fluconazole / Placebo
Started | 147 | 72
Completed | 123 | 62
Not Completed | 24 | 10
Period: 48-Week Maintenance Phase
Arm/Group | Oteseconazole (VT-1161) | Fluconazole / Placebo
Started | 123 | 62
Completed | 112 | 55
Not Completed | 11 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oteseconazole (VT-1161) | Fluconazole / Placebo | Total
Number analyzed (Participants) | 147 | 72 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.7) | 36 (11.7) | 35 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 72 | 219
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 27 | 74
  White | 88 | 42 | 130
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 147 | 72 | 219

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 1 or More Culture-verified Acute VVC Episodes During the Maintenance Phase of the Study in the Intent-to-treat (ITT) Population
Description: The primary efficacy outcome measure was the percentage of subjects with 1 or more culture-verified acute VVC episodes during the maintenance phase (post-randomization through Week 48) in the intent-to-treat population, which includes subjects who failed to clear their initial acute VVC episode during the induction phase. An acute VVC episode during the maintenance phase (considered a recurrent episode) was defined as a positive fungal culture for Candida species and a clinical signs and symptoms score of ≥3. To calculate the signs and symptoms score, each vulvovaginal sign (erythema, edema, excoriation) and symptom (itching, burning, irritation) was scored using the following scale, with a higher score indicating a worse outcome.
  0 = none (complete absence of any sign or symptom), 1 = mild (slight), 2 = moderate (definitely present), 3 = severe (marked, intense)
Time Frame: 48 Weeks
Population: Analysis was performed on the ITT population which includes subjects who failed to clear their initial acute VVC episode during the induction phase. The ITT population was defined as all randomized subjects. Missing values were imputed with multiple imputation using the following auxiliary information: treatment, baseline body mass index, baseline age, ethnicity, and visit. The 'percentage of participants' measure represents an average of 10 individual tests using multiple imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Oteseconazole (VT-1161) | Fluconazole / Placebo
Number analyzed (Participants) | 147 | 72
percentage of participants | 5.1 | 42.2

ADVERSE EVENTS:
Time Frame: Day 1 through Week 50
Description: The safety population was defined as all randomized subjects who received at least 1 dose of investigational product. Treatment-emergent adverse events were defined as adverse events that occurred after the subject received her initial dose of investigational product. One subject assigned to the oteseconazole (VT-1161) arm was not included in the safety population because she did not receive any investigation product.
Groups:
- Oteseconazole (Induction Phase): 600mg oteseconazole on Day 1 and 450mg oteseconazole on Day 2
- Oteseconazole (Maintenance Phase): 150mg oteseconazole once weekly for 11 weeks starting on Day 14.
- Fluconazole (Induction Phase): 150mg fluconazole every 72 hours in 3 sequential doses starting on Day 1
- Placebo (Maintenance Phase): Placebo once weekly for 11 weeks starting on Day 14.
Arm/Group | Oteseconazole (Induction Phase) | Oteseconazole (Maintenance Phase) | Fluconazole (Induction Phase) | Placebo (Maintenance Phase)
All-Cause Mortality (participants affected / at risk) | 0/146 | 1/123 | 0/72 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/146 | 3/123 | 0/72 | 1/62
Other Adverse Events (participants affected / at risk) | 8/146 | 35/123 | 8/72 | 21/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (Induction Phase) (N=146) | Oteseconazole (Maintenance Phase) (N=123) | Fluconazole (Induction Phase) (N=72) | Placebo (Maintenance Phase) (N=62)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (Induction Phase) (N=146) | Oteseconazole (Maintenance Phase) (N=123) | Fluconazole (Induction Phase) (N=72) | Placebo (Maintenance Phase) (N=62)
Urinary tract infection (Infections and infestations) | 1 (1) | 17 (21) | 3 (3) | 11 (11)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 16 (24) | 2 (2) | 9 (15)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 7 (8) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Fungal infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 2 (4)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 5 (5) | 2 (2) | 4 (10)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 6 (7) | 0 (0) | 3 (5)
Fatigue (General disorders) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither institution nor investigator can disclose information pertaining to study until sponsor issues multi-center publication. If multi-center publication is not issued within 18 months of study completion and database lock at all sites, sponsor has 30 days from receipt to review institution's and/or investigator's communication and can require removal of confidential information other than study data and/or delay release of institution's and/or investigator's communication for 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT03840616/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03840616/SAP_001.pdf